CLINICAL TRIAL: NCT04500132
Title: Phase 2, Multi-center, Randomized, Double-blind, Placebo- Controlled Study to Evaluate the Safety and Efficacy of EC-18 in COVID-19 Infection to Pneumonia
Brief Title: To Evaluate Safety and Efficacy of EC-18 in COVID-19 Infection to Pneumonia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Enzychem Lifesciences Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EC-18-C201
Record Dates: First submitted 2020-08-04; First posted 2020-08-05 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-02

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EC-18 Arm (Experimental): EC-18 QD
  Interventions: Drug: EC-18
- Placebo Arm (Placebo Comparator): Placebo EC-18 QD
  Interventions: Drug: Placebo EC-18

INTERVENTIONS:
Drug: EC-18 — EC-18 QD
  Arms: EC-18 Arm
Drug: Placebo EC-18 — Placebo EC-18 QD
  Arms: Placebo Arm

SUMMARY:
Prevention of COVID-19 infection to severe pneumonea or ARDS

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Male or female age 19 years or older
* Pathologically confirmed diagnosis of COVID-19 Infection to Pneumonia

Exclusion Criteria:

* Pathologically confirmed diagnosis of bacterial pneumonia or viral pneumonia
* Pregnant or nursing at the time of signing informed consent
* Known sensitivity to any study medication
* Unwilling or unable to complete study diary
* Any other condition or prior therapy that, in the opinion of the Investigator, would make the subject unsuitable for the study or unable to comply with the protocol

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2020-05-28 (Actual); Primary Completion 2021-02-04 (Actual); Study Completion 2021-02-15 (Actual)

PRIMARY OUTCOMES:
Rate of transition to ARDS | 14 days after starting IP administration

CONTACTS AND LOCATIONS:
Overall Officials: Hyewon Jeong, Principal Investigator — Chungbuk National University Hospital
Locations (1):
- Chungbuk National University Hospital, Cheongju-si, South Korea

IPD SHARING:
Plan to Share IPD: No